CLINICAL TRIAL: NCT02541110
Title: Second Trimester Maternal Serum Homocysteine Level & Uterine Artery Doppler for Prediction of Preeclampsia , Intra-Uterine Growth Retardation (IUGR) & Other Obstetric Complications
Brief Title: Prediction of Preeclampsia & Other Obstetric Complications by Serum Homocysteine & Doppler
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, suzy abdelaziz Abdelhamid, lecturer of Obgyn, Kasr El Aini Hospital
Other Study IDs: Obgyn. .
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-08

CONDITIONS: Preeclampsia; IUGR
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Second trimester homocysteine & uterine artery doppler will be assessed& the cases will be followed up till delivery for development of preeclampsia, IUGR(intra-uterine growth retardation) & other obstetric complications.

DETAILED DESCRIPTION:
Spontaneous pregnancies with no risk factors will be included. Fasting plasma total homocysteine level samples will be collected between 15th & 19th weeks.

Uterine artery doppler between 18th & 22nd weeks.

Method 1: Screen positive cases will be considered if homocysteine level above 6.3umol/l

Method 2: Screen positive cases will be considered if they had bilateral notches and a mean resistivity index (RI) above 0.55, or unilateral notches and a mean RI above 0.65, or absence of notches and a mean RI above 0.7.

Method 3: Screen positive cases will be considered if they had bilateral notches and a mean RI above 0.55, or unilateral notches and a mean RI above 0.65, or absence of notches and a mean RI above 0.7 combined with homocysteine cut off value of 6.3umol / l.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous pregnancies with no risk factors

Exclusion Criteria:

* multiple pregnancies
* non intact renal function
* hypertension
* diabetes
* folic acid supplements
* antifolate drugs

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Spontaneous pregnancies with no risk factors
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Number of pregnants who developed preeclampsia, those who developed IUGR alone and those who developed other obstetric complications as preterm labour and placental abruption | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: suzy abdelaziz, M.D., Principal Investigator — kasrelaini hospital